CLINICAL TRIAL: NCT00147511
Title: Time To Efficacy and Onset Of Action Of Linezolid In Skin and Soft Tissue Infections
Brief Title: Time To Efficacy and Onset Of Action Of Linezolid
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OXAA-0026-162
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2011-05-10 (Estimated); Status verified 2011-05

CONDITIONS: Gram-Positive Bacterial Infections; Skin and Connective Tissue Diseases
MeSH Terms: conditions — Gram-Positive Bacterial Infections; Skin and Connective Tissue Diseases | interventions — Linezolid

INTERVENTIONS:
Drug: linezolid

SUMMARY:
To assess the onset of action of linezolid

ELIGIBILITY:
Inclusion Criteria:

* suspected grampositive infection
* fever > 38 C

Exclusion Criteria:

* Infections to be treated successfully by surgical procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2003-06; Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Time to defervescence

SECONDARY OUTCOMES:
Reduction of CRP levels Reduction of leucocyte count

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer